CLINICAL TRIAL: NCT05225779
Title: A Prospective Randomized Comparison of the Effects of Sevoflurane and Desflurane Anesthesia on QT Interval Measured With Cardiac Electrophysiological Balance Index
Brief Title: The Effects of Sevoflurane and Desflurane on QT Interval Measured With Cardiac Electrophysiological Balance Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Işıl Karabeyoğlu, principal investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: E1-21-2256
Record Dates: First submitted 2022-01-05; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Sevoflurane; Desflurane; QT Interval; Electrophysiological Balance Index

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane (Active Comparator): General Anesthesia procedure with sevoflurane
  Interventions: Diagnostic Test: 12- derivation Electrocardiography
- desflurane (Active Comparator): General Anesthesia procedure with desflurane
  Interventions: Diagnostic Test: 12- derivation Electrocardiography

INTERVENTIONS:
Diagnostic Test: 12- derivation Electrocardiography — 6 precordial and 4 extremity electrodes will be placed at appropriate anatomical points and a total of 6 12-lead ECGs will be taken at different anesthesia depths before anesthesia induction and throughout the operation.

SUMMARY:
The primary aim of this study is to compare the effects of sevoflurane and desflurane on the QT interval. The secondary aim of this study is to compare the effects of drugs used in the induction and maintenance of anesthesia on the QT interval by calculating the Bazzet formula and iCEB.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II-III risk group
2. the operation time is longer than 1 hour in the Urology department.

Exclusion Criteria:

1. bundle branch block in preoperative ECG,
2. Non-sinus heart rhythm,
3. QT length in preoperative ECG,
4. using drugs that cause known QT prolongation ( beta-blocker drugs using will be included),
5. development of malignant arrhythmia that will disrupt hemodynamics in the intraoperative period,
6. patients with electrolyte disorders,
7. patient refusal -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
QTc T0 | Baseline, preoperative
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).
QTc T1 | During surgery (at the time of the anesthesia induction)
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).
QTc T2 | During surgery (at the time of MAC reached 0,6)
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).When the mac value reaches 0,6, it will be calculated from the ECG.
QTc T3 | During surgery (at the time of MAC reached1)
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).When the mac value reaches 1, it will be calculated from the ECG.
QTc T4 | During surgery (at the time of MAC reached 1,3)
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).When the mac value reaches 1,3 , it will be calculated from the ECG.
QTc T5 | During surgery (at the time of MAC reduced 0,3)
  QTc; It is calculated by dividing the QT interval by the square root of the RR interval (QTc= QT/ √RR).When the mac value reduces 0,3, it will be calculated from the ECG.
iCEB T0 | Baseline, preoperative
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS)
iCEB T1 | During surgery (at the time of the anesthesia induction)
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS)
iCEB T2 | During surgery (at the time of MAC reached 0,6)
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS) the mac value reaches 0,6, it will be calculated from the ECG.
iCEB T3 | During surgery (at the time of MAC reached 1)
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS) the mac value reaches 1, it will be calculated from the ECG.
iCEB T4 | During surgery (at the time of MAC reached 1,3)
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS) the mac value reaches 1,3, it will be calculated from the ECG.
iCEB T5 | During surgery (at the time of MAC reduced 0,3)
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS) when the mac value reduces 0,3, it will be calculated from the ECG.

CONTACTS AND LOCATIONS:
Overall Officials: ışıl karabeyoğlu, Principal Investigator — ankara ch bilkent; betül güven aytaç, Study Chair — Ankara CH bilkent

IPD SHARING:
Plan to Share IPD: No